CLINICAL TRIAL: NCT05741151
Title: Evaluation of Peripheral Catecholaminergic System in Neurodegenerative Diseases of the Central Nervous System. A Pilot Study.
Brief Title: Superior Cervical Ganglion in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4656
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: Superior Cervical Ganglion; Catecholaminergic system; Neurodegeneration; Neuroregeneration
MeSH Terms: conditions — Parkinson Disease; Nerve Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET-Neck Parkinsonian patients (Experimental): Brain and neck PET-CT with 68Ga-PSMA scan would be administered
  Interventions: Diagnostic Test: PET-Neck Parkinsonian patients

INTERVENTIONS:
Diagnostic Test: PET-Neck Parkinsonian patients — Brain and neck PET-CT scan with 68Ga-PSMA to detect metabolism in the Superior Cervical Ganglion of both sides.

SUMMARY:
In several neurodegenerative diseases, such as Parkinson's disease, the progressive loss of neurons of monoaminergic systems leads to the development of characteristic clinical manifestations.

Therefore, since the discovery that neurodegenerative phenomena are the basis of these Central Nervous System (CNS) diseases, re-innervation strategies have been studied that would allow to stop or at least slow down neurodegenerative phenomena, restoring lost catecholaminergic transmission.

Cell therapy in Parkinson's disease aims to treat motor disorders, but should not affect cognitive disorders that result from pathological alterations external to CNS and affecting other transmission systems, such as noradrenergic and cholinergic. These limitations lead to the search for new approaches based on the use of different cell types, but currently these scenarios still seem far away.

The theme of cerebral re-innervation in the treatment of neurodegenerative diseases is at the center of numerous translational and clinical research studies, developed according to various approaches and models, which testify to all the complexity and charm of the subject. Among the possible sources for a catecholamine reinnervation in Parkinson's disease, Superior Cervical Ganglion (SCG) could represent a valid autologous source: however, there is no functional evaluation in the literature that expresses the involvement or not of the ganglion in the neurodegenerative process.

This clinical study project is the first and essential phase of a larger project aimed at verifying the possibility of autologous catecholamine reinnervation in degenerative diseases of the CNS using the peripheral catecholamine system and in particular the superior cervical ganglion (GCS).

The aim of this project is to evaluate whether the peripheral catecholaminergic system, and in particular the SCG, is involved in the process of neurodegeneration. For this purpose, for an "in vivo" functional study, the suitability of the PET-CT 68Ga-PSMA examination will be studied in particular.

DETAILED DESCRIPTION:
1. (visit 1) The multidisciplinary team (neurologist, neuroradiologist, nuclear doctor and neurosurgeon) illustrates the research project to the patient eligible for the study: in case of consent to participation, informed consent is signed
2. (visit 2) Review of inclusion and exclusion criteria. Neurological evaluation Patients will undergo a complete neurological examination by a neurologist experienced in movement disorders. The inclusion criteria for this study will be verified, including the correctness of the diagnosis according to the MDS diagnostic criteria. The stage of the disease will be quantified with staging according to Hoehn and Yahr. Motor symptoms, the impact of the disease on activities of daily living, neuropsychiatric disorders and the possible presence of motor fluctuations will be quantified with the Unified Parkinson's Disease Rating scale, part I, II, III and IV. In addition, patients will be evaluated with the Mini mental Status Evaluation for cognitive impairment screening.

   The neurological evaluation will be performed a maximum of three months after the imaging examinations. Neurological evaluation will also be performed on patients in the control group, in order to exclude a diagnosis of PD.
3. (visit 3) Neuroradiology The craniocervical MRI protocol includes the sequences: axial T2 and T1 FSE/TSE, coronal T2 FSE/TSE with adipose signal saturation, axial T1 FSE/SE pre- and post-contrast (standard dose of paramagnetic MDC), 3D isotropic T1 with fat saturation, axial DWI (b 0-1000).

   The acquisition thicknesses will not exceed 3mm with a gap of 10%. 3D-STIR sequences will also be used on the 3T.

   MRI examination will be performed only on patients in the PD group.
4. (visit 4) Nuclear medicine Prostate-specific membrane antigen (PSMA) or glutamate carboxypeptidase II (GCII) is a membrane glycoprotein expressed 100-1000 times more by prostate cancer cells than by other tissues (including benign prostate tissue): its expression increases with increasing stage and grading, and in tumors resistant to antiandrogenic hormone therapy (CRPC). This makes PSMA an ideal target for detecting cancer cells with Positron Emission Tomography (PET). This method is valid in the initial staging of prostate cancer, in the re-evaluation after biochemical recurrence and in the evaluation of the response to treatment. In addition, other non-prostatic malignancies (urothelial carcinoma, bronchial carcinoma, glioblastoma), benign tumors (schwannomas, thyroid adenomas and subcutaneous or vertebral hemangiomas) as well as non-neoplastic tissues (renal tubules, duodenum, colon) have been identified by PET with 68Ga-PSMA by virtue of GCII expression.

Similarly, radiopharmaceutical uptake for PSMA has also been found in celiac, cervicothoracic (stellate) and sacral sympathetic ganglia. Histological studies have demonstrated increased GCII expression by non-myelin Schwann cells of the sympathetic nervous system ganglia . Rather limited in the literature are the studies that have analyzed the physiological greed of 68Ga-PSMA by celiac, stellate and sacral ganglia, as a potential cause of false positive findings on multimodal PET/CT or PET-MR imagin. Moreover, the uptake of 68Ga-PSMA in the superior cervical ganglion (GCS) has been analyzed only in very recent times [1].

In the present study, PET-CT imaging with 68Ga-PSMA will be used to assess the extent to which GCS uptake radiopharmaceutical for PSMA in Parkinson's disease patients. The exam will be performed at the PET Center of the Fondazione Policlinico Universitario Agostino Gemelli-IRCCS, Rome. The acquisition of the study will be performed by PET-CT tomograph 80 minutes after the administration of 68Ga-PSMA. The PET images will be evaluated independently by two Nuclear Physicians, after fusion with the MRI images for the correct anatomical localization of the GCS. After a preliminary qualitative (visual) analysis of the radiopharmaceutical uptake, a semi-quantitative evaluation will be carried out by positioning the Volume of Interest (VOI) on each of the GCS in order to calculate the Standardized Uptake Value (SUVmax). These values will be compared with those obtained in patients with prostate cancer undergoing PET-CT with 68Ga-PSMA at the same Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected with Parkinson Disease according to the criteria defined by the Movements Disorder Society

Exclusion Criteria:

* Unambiguous cerebellar abnormalities, such as cerebellar gait, limb ataxia, or cerebellar oculomotor abnormalities (eg, sustained gaze-evoked nystagmus, square wave macro jerks, hypermetric saccades)
* Palsy of vertical descending supranuclear gaze or selective slowing of vertical descending saccades
* Diagnosis of probable behavioral variant of frontotemporal dementia or primary progressive aphasia, defined according to consensus criteria, within the first 5 years of the disease
* Parkinsonian features limited to the lower limbs for more than 3 years
* Treatment with a dopamine receptor blocker or dopamine-reducing agent at a dose and time consistent with drug-induced parkinsonism
* Absence of observable response to high-dose levodopa despite at least moderate disease severity
* Unequivocal cortical sensory deficit (i.e., graphesthesia, stereognosis with intact primary sensitivities), clear ideomotor apraxia of limbs, or progressive aphasia
* Normal functional neuroimaging of the presynaptic dopaminergic system
* Documentation of an alternative condition known to induce parkinsonism and plausibly related to the patient's symptoms, or, expert medical opinion that, based on the full diagnostic evaluation, believes that an alternative syndrome is more likely than Parkinson Disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Capacity of the Superior Cervical Ganglion in parkinsonian patients | through study completion, an average of 3 years
  The capacity of the Ganglion would be assessed through the analysis of degree of captation (68Ga-CTPET)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

REFERENCES:
- [Result] Bialek EJ, Malkowski B. Are superior cervical sympathetic ganglia avid on whole body 68Ga-PSMA-11 PET/magnetic resonance?: a comprehensive morphologic and molecular assessment in patients with prostate cancer. Nucl Med Commun. 2019 Nov;40(11):1105-1111. doi: 10.1097/MNM.0000000000001083. PMID 31469805